CLINICAL TRIAL: NCT05931549
Title: Cortisol Level and Associations to Depression, Anxiety, Disease Severity and Hippocampal and Insula Volume in Anorexia Nervosa.
Brief Title: Cortisol, Hippocampus, and Insula in Anorexia Nervosa.
Acronym: EXCENTRICCAN
Status: Recruiting | Type: Observational
Sponsor: Odense University Hospital (Other)
Collaborators: Ruhr University of Bochum (Other); Umeå University (Other)
Responsible Party: Sponsor
Other Study IDs: EXCENTRICCAN
Record Dates: First submitted 2023-02-20; First posted 2023-07-05 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2024-02

CONDITIONS: Anorexia Nervosa; Stress
Keywords: anorexia nervosa; Cortisol; Insula; Hippocampus
MeSH Terms: conditions — Anorexia Nervosa

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples Without DNA — Blood, saliva, urine, hair
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients in treatment for severe anorexia nervosa: Treatment as usual.
- Age matched healthy controls: No treatment.

SUMMARY:
EXCENTRICC is a platform for scientific collaboration between different disciplines, all working on a common theme: adrenocortical hormones. In this EXCENTRICC sub-study, associations are studied between cortisol levels and depression, anxiety, disease severity and hippocampal and insula volume in the brain in anorexia nervosa.

DETAILED DESCRIPTION:
Anorexia nervosa, cortisol, hippocampus, and insula Anorexia nervosa (AN) erodes quality of life, carries the highest fatality rate of any psychiatric disease and any other chronic disease in adolescence, and poses a huge health economic burden. There has been no significant improvement of treatments since the disease was described in the last century, and only a few pharmacologic treatments have been tested in a limited number of small, controlled studies. However, weight restoration is associated with cognitive improvements.

Starvation as well as psychological stress activates the hypothalamic - pituitary - adrenal (HPA) axis with secondary anorectic, depressiogenic, and cognition-impairing effects. It has been observed that the cortisol level correlated positively with anxiety and depression in AN. Thus, glucocorticoids may be involved in a vicious circle in the development and maintenance of AN.

The hippocampus in the limbic system contains glucocorticoid receptors and is a critical structure for emotional processes as well as memory functions. Hippocampal atrophy clearly has been related to chronic stress and hypercortisolemia in studies on Cushing´s syndrome, depression and AN. However, the cause - effect associations need to be resolved by further biochemical and neuroimaging experimental studies. Compared to other mental health disorders, the number of neuroimaging studies in AN is relatively small. However, studies have revealed global and regional grey matter volume reduction as well as white matter microstructure alterations. A meta-analysis showed that adolescent patients had greater reduction in grey matter volume than adults. Other affected neuroanatomic regions are the prefrontal, parietal and temporal cortex, amygdala, insula, thalamus and cerebellum as well as various white matter tracts such as corona radiata and superior longitudinal fascicules. Structural and functional alterations have been detected in the early course of the disease, most of them being partially or totally reversible with weight restoration. An area of high interest is the insula. The insular cortex is implicated in a variety of functions such as emotional awareness, decision-making and complex social functions like empathy. An additional key function of the insula is the integration of interoceptive information, i.e., internal physical sensations including hunger. Furthermore, the right insula specifically is involved in "self-recognition". MRI studies have revealed increased volume of the right insula in adolescent and adult patients with AN and this finding has been correlated with the rumination of being fat while being emaciated.

Cortisol synthesis inhibition Preliminary experimental evidence indicate that inhibition of pharmacological cortisol synthesis may have therapeutic effects on depression. Mifepristone is a competitive cortisol antagonist used therapeutically in Cushing's syndrome. The elimination half-life is approximately 20 h. In a Cochrane metanalysis of treatment with anti-glucocorticoid drugs for psychosis and major depression, it was concluded that mifepristone in a dose range of 600-1200 mg/day may ameliorate psychotic and depressive symptoms in patients with major depression. In four small studies, the incidence of side effects of mifepristone was similar to the placebo groups. The effect of mifepristone in AN has only been explored in one study with eight patients in a single dose of 10 mg/kg which demonstrated increase in urinary free cortisol excretion and in early morning cortisol plasma levels.

Cortisol assessments In healthy subjects, circulating cortisol has a diurnal pattern, with a stable day-night-sleep rhythm. Cortisol levels reach maximum concentrations in the morning and nadir at midnight. In plasma, cortisol circulates in three fractions: 80% circulates bound to cortisol binding globulin (CBG), 10-15% is bound to albumin, whereas the remaining 5-10% circulates as free and biologically active cortisol. Estrogens stimulate CBG during treatment with oral contraception (OC) which leads to elevated total cortisol concentrations. Conversely, in severe illness, the stress imposed upon the patient causes CBG to decrease (mediated by interleukin-6 levels) which results in low total plasma cortisol levels. The HPA-axis activity may be assessed by measuring cortisol in plasma, saliva, urine, and hair. Urine, saliva and hair cortisol represent the free forms of cortisol, but most saliva assays do not take the rapid conversion of cortisol to cortisone into account, and further, saliva concentrations may be biased by traces of oral medications and smoking. Furthermore, there are advantages and drawbacks of acute assessment of cortisol (serum or saliva) versus integrated cortisol levels (diurnal urine or hair cortisol). The steroid metabolic pathway is extremely complicated and a detailed "foot-print" of steroid metabolites may potentially add information beyond that of cortisol measurement. For instance, a ratio between different down-stream metabolites of cortisol may provide information about the course of cortisol excess. Finally, FK506-binding immunophilins, Fkbp4 and Fkbp5 regulate nuclear translocation of the glucocorticoid receptor, resulting in modulation of the glucocorticoid action. Measuring methylation status of the FKBP5 gene in leukocytes are suggested to be a biomarker for Glucocorticoid Replacement.

Aim and perspectives The study will provide novel, original data, and insight into the pathogenetic role of cortisol, hippocampal and insular volume in severe AN. This insight may potentially generate highly warranted new therapeutic targets.

Hypothesis and research questions

1. It is hypothesized that cortisol levels assessed by mean concentrations in plasma, saliva, urine, and hair are associated with depression, anxiety, and severity of AN, assessed based on validated psychometric measures, degree of underweight, and impairment of disease-specific HRQOL in AN.
2. It is hypothesized that cortisol levels are associated with altered volumes of hippocampus and insula assessed by MRI.
3. The above-mentioned associations are hypothesized to be significantly stronger for unbound cortisol concentrations than that for traditional total concentration in plasma. Thus, free unbound cortisol may prove to have the potential to be a clinically useful state-related biomarker in AN.

ELIGIBILITY:
Inclusion Criteria:

1. Women who fulfill the criteria for AN according to the Diagnostic and Statistical Manual of Mental Disorders (DSM), version 5 (APA, 2013).
2. BMI < 16.

Exclusion Criteria:

1. Current treatment with glucocorticoids.
2. Current use of oral contraceptives.
3. Unstable acute somatic comorbidity, e.g., infection.
4. Any kind of metal prostheses or -implants.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — The disease anorexia nervosa is predominantly observed in women (approximately 95%).
Study Population: Women with anorexia nervosa, treatment seeking at Center for Eating Disorders at Odense University Hospital or via advertising on social media.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Hippocampus total volumen (cm3) | Cross sectional (AN patients during a treatment course)
  MRI
Insula total volumen (cm3) | (AN patients during a treatment course)
  MRI
Plasma cortisol level (mmol/l) | AN patients during a treatment course at any time in relation to the duration of the illness and course of treatment.
Cortisol diurnal excretion (nmol/d) | AN patients during a treatment course at any time in relation to the duration of the illness and course of treatment.

SECONDARY OUTCOMES:
Symptom severity | AN patients during a treatment course at any time in relation to the duration of the illness and course of treatment.
  Eating Disorder Inventory (EDI)-3. Score 91 - 546. High score indicates high disease severity. Severity of eating disorder symptomatology will be assessed using the EDI-3. It consists of 91 items and has 11 subscales: Drive for Thinness, Bulimia, Body Dissatisfaction, Ineffectiveness, Perfectionism, Interpersonal Distrust, Introspective Awareness, Maturity Fears, Asceticism, Impulse Regulation, and Social Insecurity. Answers are given on a 6-point likert scale. The higher the score, the greater the manifestation of the trait in question. The instrument has been validated in Danish.
Depression | AN patients during a treatment course at any time in relation to the duration of the illness and course of treatment.
  Beck Depression Inventory version 2 (BDI-II). Score 0-63, high score indicates more severe symptoms of depression. BDI-II is a self-report questionnaire consisting of 21 statements that is frequently used to detect varying degrees of depression and examines symptoms such as loss of joy, sadness and guilt, as well as physical symptoms, including energy loss, altered appetite, difficulty concentrating, and fatigue / exhaustion. Answers are given in relation to how well the described symptom describes one's thoughts, feelings, and behavior over the past two weeks. Answers are scored from 0-3. The BDI has shown high internal consistency and has been validated for eating disorders.
Anxiety | AN patients during a treatment course at any time in relation to the duration of the illness and course of treatment.
  Hospital Anxiety and Depression Scale (HADS). Score 14-70. High score indicates high symptom severity. Seven measure symptoms of anxiety and 7 measure symptoms of depression. Answers are given for the preceding week and are calculated on a 5-point scale.
Quality of life | AN patients during a treatment course at any time in relation to the duration of the illness and course of treatment.
  Disease specific health-related quality of life in eating disorders (EDQLS). Score 40-200. High score indicates high health-related quality of life. The term health-related quality of life (HRQoL) is used to refer to quality of life aspects related to ill-health, disability, and treatment and is a multidimensional concept that describes physical, social, and psychological well-being and functioning. Patient-reported HRQoL is particularly relevant in anorexia nervosa due to the ego-syntonic nature of the disease, and its omission this may lead to large discrepancies between what the patient experiences and what the clinician perceives. EDQLS was developed and validated in both clinical and non-clinical settings and is available in.

CONTACTS AND LOCATIONS:
Overall Officials: René K Støving, PhD, Principal Investigator — Odense University Hospital
Locations (1):
- Odense University Hospital, Odense, Denmark

IPD SHARING:
Plan to Share IPD: No